CLINICAL TRIAL: NCT05428436
Title: Relative Bioavailability Comparison of BI 1015550 as the Intended Commercial Formulation (iCF) Versus Trial Formulation 2 and iCF With and Without Food Following Oral Administration in Healthy Subjects (an Open-label, Randomised, Single-dose, Three-way Crossover Trial)
Brief Title: A Study in Healthy People to Compare 2 Different Formulations of BI 1015550 Taken With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0028; 2021-006890-44 (EudraCT Number)
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- R/T1/T2 (Experimental): Three period crossover with treatments in the following order:
  Reference (R): three 6 milligram BI 1015550 film-coated tablets of Trial Formulation 2 (TF2) taken orally following an overnight fast of at least 10 hours.
  Test treatment 1 (T1): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following an overnight fast of at least 10 hours.
  Test treatment 2 (T2): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following a high-calorie breakfast.
  Periods were separated by a washout period of at least 7 days between treatments.
  Interventions: Drug: Reference (R); Drug: Test treatment 1 (T1); Drug: Test treatment 2 (T2)
- T1/T2/R (Experimental): Three period crossover with treatments in the following order:
  Test treatment 1 (T1): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following an overnight fast of at least 10 hours.
  Test treatment 2 (T2): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following a high-calorie breakfast.
  Reference (R): three 6 milligram BI 1015550 film-coated tablets of Trial Formulation 2 (TF2) taken orally following an overnight fast of at least 10 hours.
  Periods were separated by a washout period of at least 7 days between treatments.
  Interventions: Drug: Reference (R); Drug: Test treatment 1 (T1); Drug: Test treatment 2 (T2)
- T2/R/T1 (Experimental): Three period crossover with treatments in the following order:
  Test treatment 2 (T2): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following a high-calorie breakfast.
  Reference (R): three 6 milligram BI 1015550 film-coated tablets of Trial Formulation 2 (TF2) taken orally following an overnight fast of at least 10 hours.
  Test treatment 1 (T1): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following an overnight fast of at least 10 hours.
  Periods were separated by a washout period of at least 7 days between treatments
  Interventions: Drug: Reference (R); Drug: Test treatment 1 (T1); Drug: Test treatment 2 (T2)

INTERVENTIONS:
Drug: Reference (R) — Reference (R): three 6 milligram BI 1015550 film-coated tablets of Trial Formulation 2 (TF2) taken orally following an overnight fast of at least 10 hours.
  Other Names: Nerandomilast; JASCAYD®
Drug: Test treatment 1 (T1) — Test treatment 1 (T1): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following an overnight fast of at least 10 hours.
  Other Names: Nerandomilast; JASCAYD®
Drug: Test treatment 2 (T2) — Test treatment 2 (T2): one 18 milligram BI 1015550 film-coated tablet of the intended commercial formulation (iCF) taken orally following a high-calorie breakfast.
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 1015550 intended Commercial Formulation (iCF) compared with Trial Formulation 2 (TF2) and the effect of food on the pharmacokinetics of BI 1015550 iCF following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 55 years (inclusive).
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Council for Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Either male subject, or female subject who meet any of the following criteria from 30 days before drug administration until 7 days after trial completion:

  * Use of non-oral hormonal contraception associated with inhibition of ovulation:

intravaginal or transdermal combinations of estrogen and progestogen or injectable or implantable progestogen.

* Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).
* Sexually abstinent, i.e. complete abstinence from male-female sex when this is in line with the preferred and usual lifestyle of the study participant. Periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods; declaration of abstinence for the duration of exposure to study drug; and withdrawal are not acceptable.
* Vasectomised sexual partner with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate, provided that partner is the sole sexual partner of the study participant
* Surgically sterilised (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy, bilateral tubal occlusion).
* Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory).

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator-
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm).
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance.
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair).
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders (including but not limited to major depressive disorder or history of suicide attempts).
* History of relevant orthostatic hypotension, fainting spells, or blackouts. Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was a randomised, open-label, single-dose, three-way crossover design. The subjects were randomly allocated to 1 of 3 treatment sequences. Each subject participated in 3 treatment periods, receiving a single dose in each, with a washout period of at least 7 days between treatments.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Period 1
Arm/Group | R/T1/T2 | T1/T2/R | T2/R/T1
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Period 1 - 2 washout
Arm/Group | R/T1/T2 | T1/T2/R | T2/R/T1
Started | 8 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Period: Period 2
Arm/Group | R/T1/T2 | T1/T2/R | T2/R/T1
Started | 7 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Period 2 - 3 washout
Arm/Group | R/T1/T2 | T1/T2/R | T2/R/T1
Started | 7 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 0 | 0 | 0
Period: Period 3
Arm/Group | R/T1/T2 | T1/T2/R | T2/R/T1
Started | 7 | 8 | 8
Completed | 7 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | R/T1/T2 | T1/T2/R | T2/R/T1 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (11.3) | 40.0 (11.8) | 39.6 (14.2) | 39.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 9
  Male | 3 | 7 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 8 | 7 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: Within 3 hours before and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144 hours following drug administration.
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects who were treated with at least one dose of trial drug and who provided at least one Pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomol/Liter
Groups:
- Reference treatment (R) - fasted: Reference (R): three 6 milligram BI 1015550 film-coated tablets of Trial Formulation 2 (TF2) taken orally following an overnight fast of at least 10 hours.
- Test treatment 1 (T1) - fasted: Test treatment 1 (T1): one 18 milligram BI 1015550-film-coated tablet of the intended commercial formulation (iCF) taken orally following an overnight fast of at least 10 hours.
- Test treatment 2 (T2) - fed: Test treatment 2 (T2): one 18 milligram BI 1015550 film--coated tablet of the intended commercial formulation (iCF) taken orally following a high-calorie breakfast.
Arm/Group | Reference treatment (R) - fasted | Test treatment 1 (T1) - fasted | Test treatment 2 (T2) - fed
Number analyzed (Participants) | 24 | 23 | 23
hours*nanomol/Liter | 2290 (194) | 2740 (34.7) | 3000 (31.2)
Statistical Analysis 1: Comparison: Reference treatment (R) - fasted vs Test treatment 1 (T1) - fasted; Analysis of Variance (ANOVA) model (logarithmic scale) with the effects: sequence, subjects within sequences, period, and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; gMean ratio = 121.12, 90% CI 2-sided [86.14 to 170.30] — gMean ratio: T1/R. Intra-individual Geometric coefficient of variation [%] = 78.5
Statistical Analysis 2: Comparison: Test treatment 1 (T1) - fasted vs Test treatment 2 (T2) - fed; ANOVA model (logarithmic scale) with the effects: sequence, subjects within sequences, period, and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; gMean ratio = 108.13, 90% CI 2-sided [76.68 to 152.48] — gMean ratio: T2/T1. Intra-individual Geometric coefficient of variation [%] = 78.5

2. Primary Outcome: Area Under the Concentration-time Curve of R-BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of R-BI 1015550 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). The endpoint was analyzed additionally for the chirally pure (R) form of BI 1015550 (R-BI 1015550, the pharmacologically active form).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomol/Liter
Arm/Group | Reference treatment (R) - fasted | Test treatment 1 (T1) - fasted | Test treatment 2 (T2) - fed
Number analyzed (Participants) | 24 | 23 | 23
hours*nanomol/Liter | 1900 (197) | 2310 (29.6) | 2500 (26.9)
Statistical Analysis 1: Comparison: Reference treatment (R) - fasted vs Test treatment 1 (T1) - fasted; Analysis of Variance (ANOVA) model (logarithmic scale) with the effects: sequence, subjects within sequences, period, and treatment (restricted to the two formulation groups (T1 & R)). The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; gMean ratio = 122.01, 90% CI 2-sided [79.25 to 187.84] — gMean ratio: T1/R. Intra-individual Geometric coefficient of variation [%] = 104.0
Statistical Analysis 2: Comparison: Test treatment 1 (T1) - fasted vs Test treatment 2 (T2) - fed; ANOVA model (logarithmic scale) with the effects: sequence, subjects within sequences, period, and treatment (restricted to the two treatment groups (T1 & T2)). The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; gMean ratio = 108.56, 90% CI 2-sided [104.33 to 112.97] — gMean ratio: T2/T1. Intra-individual Geometric coefficient of variation [%] = 7.8

3. Primary Outcome: Maximum Measured Concentration of BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of BI 1015550 in plasma (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Liter
Arm/Group | Reference treatment (R) - fasted | Test treatment 1 (T1) - fasted | Test treatment 2 (T2) - fed
Number analyzed (Participants) | 24 | 23 | 23
nanomol/Liter | 313 (165) | 364 (36.6) | 323 (22.7)
Statistical Analysis 1: Comparison: Reference treatment (R) - fasted vs Test treatment 1 (T1) - fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; gMean ratio = 118.00, 90% CI 2-sided [85.82 to 162.25] — gMean ratio: T1/R. Intra-individual Geometric coefficient of variation [%] = 72.2
Statistical Analysis 2: Comparison: Test treatment 1 (T1) - fasted vs Test treatment 2 (T2) - fed; [analysis description as in outcome 1, analysis 2]; Test type: Other; gMean ratio = 87.94, 90% CI 2-sided [63.77 to 121.28] — gMean ratio: T2/T1. Intra-individual Geometric coefficient of variation [%] = 72.2

4. Primary Outcome: Maximum Measured Concentration of R-BI 1015550 in Plasma (Cmax)
Description: Maximum measured concentration of R-BI 1015550 in plasma (Cmax). The endpoint was analyzed additionally for the chirally pure (R) form of BI 1015550 (R-BI 1015550, the pharmacologically active form).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/Liter
Arm/Group | Reference treatment (R) - fasted | Test treatment 1 (T1) - fasted | Test treatment 2 (T2) - fed
Number analyzed (Participants) | 24 | 23 | 23
nanomol/Liter | 307 (166) | 352 (35.4) | 319 (23.8)
Statistical Analysis 1: Comparison: Reference treatment (R) - fasted vs Test treatment 1 (T1) - fasted; ANOVA model (logarithmic scale) with the effects: sequence, subjects within sequences, period, and treatment (restricted to the two formulation groups (T1 & R)). The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Test type: Other; gMean ratio = 115.63, 90% CI 2-sided [77.64 to 172.22] — gMean ratio: T1/R. Intra-individual Geometric coefficient of variation [%] = 93.3
Statistical Analysis 2: Comparison: Test treatment 1 (T1) - fasted vs Test treatment 2 (T2) - fed; [analysis description as in outcome 2, analysis 2]; Test type: Other; gMean ratio = 90.74, 90% CI 2-sided [80.82 to 101.87] — gMean ratio: T2/T1. Intra-individual Geometric coefficient of variation [%] = 23.0

5. Secondary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity, Predicted (AUC0-∞,Pred)
Description: Area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 extrapolated to infinity, predicted (AUC0-∞,pred).
Time Frame: as for outcome 1
Population: Pharmacokinetic parameter analysis set (PKS): This set included all subjects who were treated with at least one dose of trial drug and who provided at least one Pharmacokinetic (PK) endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Endpoint only includes subjects where AUC0-∞,pred could be calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomol/Liter
Arm/Group | Reference treatment (R) - fasted | Test treatment 1 (T1) - fasted | Test treatment 2 (T2) - fed
Number analyzed (Participants) | 23 | 23 | 23
hours*nanomol/Liter | 2970 (30.0) | 2780 (35.1) | 3050 (31.7)
Statistical Analysis 1: Comparison: Reference treatment (R) - fasted vs Test treatment 1 (T1) - fasted; [analysis description as in outcome 1, analysis 2]; Test type: Other; gMean ratio = 93.79, 90% CI 2-sided [90.49 to 97.21] — gMean ratio: T1/R. Intra-individual Geometric coefficient of variation [%] = 7.1
Statistical Analysis 2: Comparison: Test treatment 1 (T1) - fasted vs Test treatment 2 (T2) - fed; [analysis description as in outcome 1, analysis 2]; Test type: Other; gMean ratio = 109.51, 90% CI 2-sided [105.72 to 113.44] — gMean ratio: T2/T1. Intra-individual Geometric coefficient of variation [%] = 7.1

6. Secondary Outcome: Area Under the Concentration-time Curve of R-BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity, Predicted (AUC0-∞,Pred)
Description: Area under the concentration-time curve of R-BI 1015550 in plasma over the time interval from 0 extrapolated to infinity, predicted (AUC0-∞,pred). The endpoint was analyzed additionally for the chirally pure (R) form of BI 1015550 (R-BI 1015550, the pharmacologically active form).
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanomol/Liter
Arm/Group | Reference treatment (R) - fasted | Test treatment 1 (T1) - fasted | Test treatment 2 (T2) - fed
Number analyzed (Participants) | 23 | 23 | 23
hours*nanomol/Liter | 2460 (27.0) | 2340 (30.0) | 2530 (27.2)
Statistical Analysis 1: Comparison: Reference treatment (R) - fasted vs Test treatment 1 (T1) - fasted; [analysis description as in outcome 4, analysis 1]; Test type: Other; gMean ratio = 95.01, 90% CI 2-sided [91.39 to 98.77] — gMean ratio: T1/R. Intra-individual Geometric coefficient of variation [%] = 7.5
Statistical Analysis 2: Comparison: Test treatment 1 (T1) - fasted vs Test treatment 2 (T2) - fed; [analysis description as in outcome 2, analysis 2]; Test type: Other; gMean ratio = 108.30, 90% CI 2-sided [103.90 to 112.89] — gMean ratio: T2/T1. Intra-individual Geometric coefficient of variation [%] = 8.2

ADVERSE EVENTS:
Time Frame: Adverse events: From trial medication intake till the end of the residual effect period (REP), up to 7 days. All-Cause Mortality: Up to 14 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug.
Arm/Group | Reference Treatment (R) - Fasted | Test Treatment 1 (T1) - Fasted | Test Treatment 2 (T2) - Fed
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 5/24 | 3/23 | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reference Treatment (R) - Fasted (N=24) | Test Treatment 1 (T1) - Fasted (N=23) | Test Treatment 2 (T2) - Fed (N=23)
Headache (Nervous system disorders) | 5 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT05428436/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT05428436/SAP_001.pdf